CLINICAL TRIAL: NCT03076775
Title: Fetal Metabolic Consequences of Late Preterm Steroid Exposure
Brief Title: Euglycemia After Antenatal Late Preterm Steroids, the E-ALPS Study
Acronym: E-ALPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-1970; 1R03HD096188-01 (NIH)
Record Dates: First submitted 2017-03-01; First posted 2017-03-10 (Actual); Results first posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-12

CONDITIONS: Pregnancy Preterm; Neonatal Hypoglycemia; Hyperglycemia Drug Induced
Keywords: Betamethasone; Late preterm; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Women will undergo regular maternal blood glucose screening and treatment of hyperglycemia following BMZ administration to achieve maternal glycemic control until delivery or hospital discharge, for a maximum of 5 days.
  Interventions: Other: Maternal glycemic control
- Usual Care (No Intervention): Routine antenatal care will be performed without any maternal blood glucose screening nor treatment as is usual care at each of the study sites.

INTERVENTIONS:
Other: Maternal glycemic control — Maternal capillary blood glucose testing will be performed according to oral intake status: every 2 hours if not eating (NPO) or fasting and 1-hour postprandial if eating regular meals. Hyperglycemia, defined based on the American Diabetes Association and the American College of Obstetricians and Gynecologists recommendations as well as current practice at study sites, will be treated according to study guidelines based on oral intake status: insulin infusion if NPO and subcutaneous insulin if eating regular meals.
  Arms: Intervention

SUMMARY:
Annually in the U.S 300,000 neonates are born late preterm, defined as 34 weeks 0 days - 36 weeks 6 days. The Antenatal Late Preterm Steroids (ALPS) Trial demonstrated that maternal treatment with betamethasone in the late preterm period significantly reduces neonatal respiratory complications, but also increases neonatal hypoglycemia, compared to placebo.

This research study will attempt to answer the following primary question: Does a management protocol aimed at maintaining maternal euglycemia after ALPS decrease fetal hyperinsulinemia, compared to usual antepartum care?

DETAILED DESCRIPTION:
Euglycemia after Antenatal Late Preterm Steroids, the E-ALPS Study:

There is a fundamental gap in understanding the adverse metabolic effects of antenatal late preterm steroids (ALPS). In 2016, an important randomized clinical trial of 2827 late preterm pregnancies showed that antenatal betamethasone (BMZ) significantly reduced neonatal respiratory complications compared with placebo. However, those neonates exposed to BMZ were also more likely to have hypoglycemia at birth. This unexpected adverse outcome raised concern among both obstetricians and neonatologists and remains an important knowledge gap to be filled. The rationale for the proposed research is that steroid-induced maternal hyperglycemia leads to transient fetal hyperinsulinemia, which causes hypoglycemia in neonates that are delivered during this time-period. Thus, the fetal metabolic consequences and subsequent neonatal hypoglycemia observed after exposure to BMZ in utero can be prevented by achieving maternal euglycemia prior to delivery.

This protocol describes a randomized clinical trial to evaluate whether screening for and treatment of steroid-induced hyperglycemia in non-diabetic women treated with BMZ in the late preterm period can decrease the rate of fetal hyperinsulinemia, thus reducing neonatal hypoglycemia and improving short-term neonatal outcomes.

This study was formerly approved as Institutional Review Board #16-3200.

ELIGIBILITY:
Inclusion Criteria:

* Singleton gestation with no known major fetal anomalies
* Gestational age at randomization between 34 weeks 0 days and 36 weeks 5 days
* Receiving antenatal betamethasone due to high probability of delivery in late preterm period

Exclusion Criteria:

* Pre-gestational or gestational diabetes mellitus
* Maternal contraindication to insulin
* Planned outpatient treatment with antenatal betamethasone
* Participation in clinical trial that could affect primary outcome or participation in this trial in a previous pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Recruiting pregnant females
Enrollment: 86 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashley N Battarbee, MD, MSCR, Principal Investigator — University of Alabama at Birmingham; Kim Boggess, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No
Data collected as a part of this trial will only be available to the study team. Protected health information will only be available to the recruiting site in order to complete data abstraction.

REFERENCES:
- [Background] Gyamfi-Bannerman C, Thom EA, Blackwell SC, Tita AT, Reddy UM, Saade GR, Rouse DJ, McKenna DS, Clark EA, Thorp JM Jr, Chien EK, Peaceman AM, Gibbs RS, Swamy GK, Norton ME, Casey BM, Caritis SN, Tolosa JE, Sorokin Y, VanDorsten JP, Jain L; NICHD Maternal-Fetal Medicine Units Network. Antenatal Betamethasone for Women at Risk for Late Preterm Delivery. N Engl J Med. 2016 Apr 7;374(14):1311-20. doi: 10.1056/NEJMoa1516783. Epub 2016 Feb 4. PMID 26842679
- [Background] Martin JA, Hamilton BE, Osterman MJ, Driscoll AK, Mathews TJ. Births: Final Data for 2015. Natl Vital Stat Rep. 2017 Jan;66(1):1. PMID 28135188
- [Background] McIntire DD, Leveno KJ. Neonatal mortality and morbidity rates in late preterm births compared with births at term. Obstet Gynecol. 2008 Jan;111(1):35-41. doi: 10.1097/01.AOG.0000297311.33046.73. PMID 18165390
- [Background] Consortium on Safe Labor; Hibbard JU, Wilkins I, Sun L, Gregory K, Haberman S, Hoffman M, Kominiarek MA, Reddy U, Bailit J, Branch DW, Burkman R, Gonzalez Quintero VH, Hatjis CG, Landy H, Ramirez M, VanVeldhuisen P, Troendle J, Zhang J. Respiratory morbidity in late preterm births. JAMA. 2010 Jul 28;304(4):419-25. doi: 10.1001/jama.2010.1015. PMID 20664042
- [Background] Gilbert WM, Nesbitt TS, Danielsen B. The cost of prematurity: quantification by gestational age and birth weight. Obstet Gynecol. 2003 Sep;102(3):488-92. doi: 10.1016/s0029-7844(03)00617-3. PMID 12962929
- [Background] Jolley JA, Rajan PV, Petersen R, Fong A, Wing DA. Effect of antenatal betamethasone on blood glucose levels in women with and without diabetes. Diabetes Res Clin Pract. 2016 Aug;118:98-104. doi: 10.1016/j.diabres.2016.06.005. Epub 2016 Jun 17. PMID 27351800
- [Background] Langen ES, Kuperstock JL, Sung JF, Taslimi M, Byrne J, El-Sayed YY. Maternal glucose response to betamethasone administration. Am J Perinatol. 2015 Feb;30(2):143-8. doi: 10.1055/s-0034-1376387. Epub 2014 Jun 10. PMID 24915559
- [Background] Shelton SD, Boggess KA, Smith T, Herbert WN. Effect of betamethasone on maternal glucose. J Matern Fetal Neonatal Med. 2002 Sep;12(3):191-5. doi: 10.1080/jmf.12.3.191.195. PMID 12530617
- [Background] Refuerzo JS, Garg A, Rech B, Ramin SM, Vidaeff A, Blackwell SC. Continuous glucose monitoring in diabetic women following antenatal corticosteroid therapy: a pilot study. Am J Perinatol. 2012 May;29(5):335-8. doi: 10.1055/s-0031-1295642. Epub 2011 Nov 17. PMID 22094918
- [Background] Sifianou P, Thanou V, Karga H. Metabolic and hormonal effects of antenatal betamethasone after 35 weeks of gestation. J Pediatr Pharmacol Ther. 2015 Mar-Apr;20(2):138-43. doi: 10.5863/1551-6776-20.2.138. PMID 25964731
- [Background] Obenshain SS, Adam PA, King KC, Teramo K, Raivio KO, Raiha N, Schwartz R. Human fetal insulin response to sustained maternal hyperglycemia. N Engl J Med. 1970 Sep 10;283(11):566-70. doi: 10.1056/NEJM197009102831104. No abstract available. PMID 5450610
- [Background] Kuhl C, Andersen GE, Hertel J, Molsted-Pedersen L. Metabolic events in infants of diabetic mothers during first 24 hours after birth. I. Changes in plasma glucose, insulin and glucagon. Acta Paediatr Scand. 1982 Jan;71(1):19-25. doi: 10.1111/j.1651-2227.1982.tb09366.x. PMID 6753468
- [Background] American College of Obstetricians and Gynecologists' Committee on Obstetric Practice; Society for Maternal- Fetal Medicine. Committee Opinion No.677: Antenatal Corticosteroid Therapy for Fetal Maturation. Obstet Gynecol. 2016 Oct;128(4):e187-94. doi: 10.1097/AOG.0000000000001715. PMID 27661658
- [Background] Society for Maternal-Fetal Medicine (SMFM) Publications Committee. Implementation of the use of antenatal corticosteroids in the late preterm birth period in women at risk for preterm delivery. Am J Obstet Gynecol. 2016 Aug;215(2):B13-5. doi: 10.1016/j.ajog.2016.03.013. Epub 2016 Mar 15. No abstract available. PMID 26992737
- [Background] ACOG Committee on Practice Bulletins. ACOG Practice Bulletin. Clinical Management Guidelines for Obstetrician-Gynecologists. Number 60, March 2005. Pregestational diabetes mellitus. Obstet Gynecol. 2005 Mar;105(3):675-85. doi: 10.1097/00006250-200503000-00049. No abstract available. PMID 15738045
- [Background] American Diabetes Association. Standards of medical care in diabetes - 2016. Diabetes Care. 2016; 39(suppl1):S1-S106.
- [Derived] Battarbee AN, Ye Y, Szychowski JM, Casey BM, Tita AT, Boggess KA. Euglycemia after antenatal late preterm steroids: a multicenter, randomized controlled trial. Am J Obstet Gynecol MFM. 2022 Jul;4(4):100625. doi: 10.1016/j.ajogmf.2022.100625. Epub 2022 Mar 26. PMID 35346889

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Women will undergo regular maternal blood glucose screening and treatment of hyperglycemia following Betamethasone (BMZ) administration to achieve maternal glycemic control until delivery or hospital discharge, for a maximum of 5 days.
  Maternal glycemic control: Maternal capillary blood glucose testing will be performed according to oral intake status: every 2 hours if not eating (NPO) or fasting and 1-hour postprandial if eating regular meals. Hyperglycemia, defined based on the American Diabetes Association and the American College of Obstetricians and Gynecologists recommendations as well as current practice at study sites, will be treated according to study guidelines based on oral intake status: insulin infusion if NPO and subcutaneous insulin if eating regular meals.
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 44 | 42
Neonates Born During Study | 43 | 42
Umbilical Cord Blood Collected | 33 | 38
Completed | 43 | 42
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 43 | 42 | 85
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [21 to 32] | 28 [23 to 33] | 28 [22 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 42 | 85
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data unreported by 1 participant
  Participants
    Non-Hispanic Black: number analyzed (Participants) | 42 | 42 | 84
    Non-Hispanic Black | 17 | 16 | 33
    Non-Hispanic White: number analyzed (Participants) | 42 | 42 | 84
    Non-Hispanic White | 17 | 18 | 35
    Hispanic: number analyzed (Participants) | 42 | 42 | 84
    Hispanic | 8 | 7 | 15
    Other: number analyzed (Participants) | 42 | 42 | 84
    Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 42 | 85

OUTCOME MEASURES:

1. Primary Outcome: Umbilical Cord Blood C-peptide
Description: C-peptide level (ng/mL) as measure of fetal hyperinsulinemia
Time Frame: At delivery
Population: Umbilical cord blood specimen only available for 70 neonates
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Neonates Born to Mothers Receiving Intervention: Neonates born to mothers who received intervention
- Neonates Born to Mothers Receiving Usual Care: Neonates born to mothers who received usual care
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 33 | 37
ng/mL | 1.02 [0.52 to 1.86] | 1.09 [0.61 to 1.65]
Statistical Analysis 1: Comparison: Neonates Born to Mothers Receiving Intervention vs Neonates Born to Mothers Receiving Usual Care; Test type: Superiority; p = 0.97, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Umbilical Cord Blood Cortisol
Description: Cortisol level (ug/mL) as measure of fetal immune suppression
Time Frame: At delivery
Population: Umbilical cord blood specimen only available for 70 neonates
Measure: Median (Inter-Quartile Range); unit: ug/mL
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 33 | 37
ug/mL | 2.0 [1.1 to 5.1] | 2.5 [1.7 to 5.9]
Statistical Analysis 1: Comparison: Neonates Born to Mothers Receiving Intervention vs Neonates Born to Mothers Receiving Usual Care; Test type: Superiority; p = 0.24, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Umbilical Insulin-Like Growth Factor 1
Description: Insulin-like growth factor 1 level (ng/mL) as a measure of in utero metabolic status
Time Frame: At delivery
Population: Umbilical cord blood specimen only available for 71 neonates
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 33 | 38
ng/mL | 78 [53 to 98] | 58 [42 to 90]
Statistical Analysis 1: Comparison: Neonates Born to Mothers Receiving Intervention vs Neonates Born to Mothers Receiving Usual Care; Test type: Superiority; p = 0.15, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Umbilical Cord Blood Leptin
Description: Leptin level (ng/mL) as measure of fetal adiposity
Time Frame: At delivery
Population: Umbilical cord blood specimen only available for 71 neonates
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 33 | 38
ng/mL | 7.5 [4.4 to 11.2] | 5.6 [3.2 to 12.6]
Statistical Analysis 1: Comparison: Neonates Born to Mothers Receiving Intervention vs Neonates Born to Mothers Receiving Usual Care; Test type: Superiority; p = 0.55, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Neonatal Hypoglycemia
Description: Number of neonates with capillary blood glucose < 40 mg/dL
Time Frame: After birth, up to 48 hours of life
Population: Glucose only available for 82 neonates
Measure: Count of Participants; unit: Participants
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 41 | 41
Participants | 20 | 21
Statistical Analysis 1: Comparison: Neonates Born to Mothers Receiving Intervention vs Neonates Born to Mothers Receiving Usual Care; Test type: Superiority; p = 0.83, Chi-squared

6. Secondary Outcome: Neonatal Hypoglycemia Treatment
Description: Number of neonates with hypoglycemia requiring treatment with dextrose gel or dextrose intravenous fluids
Time Frame: After birth, during hospital admission, assessed up to 28 days
Population: Glucose only available for 82 neonates
Measure: Count of Participants; unit: Participants
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 41 | 41
Participants | 9 | 8
Statistical Analysis 1: Comparison: Neonates Born to Mothers Receiving Intervention vs Neonates Born to Mothers Receiving Usual Care; Test type: Superiority; p = 0.79, Chi-squared

7. Secondary Outcome: Neonatal Glucose Nadir
Description: Lowest neonatal capillary blood glucose (mg/dL)
Time Frame: After birth, during hospital admission, assessed up to 28 days
Population: Glucose only available on 82 neonates
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 41 | 41
mg/dL | 42.3 (2.9) | 42.2 (2.2)
Statistical Analysis 1: Comparison: Neonates Born to Mothers Receiving Intervention vs Neonates Born to Mothers Receiving Usual Care; Test type: Superiority; p = 0.97, t-test, 2 sided

8. Secondary Outcome: Timing of Neonatal Blood Glucose Nadir
Description: Number of hours after birth when lowest neonatal capillary blood glucose was measured
Time Frame: After birth, during hospital admission, assessed up to 28 days
Population: Glucose only available on 82 neonates
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 41 | 41
hours | 1.7 [1.5 to 4.3] | 1.7 [1.4 to 3.6]
Statistical Analysis 1: Comparison: Neonates Born to Mothers Receiving Intervention vs Neonates Born to Mothers Receiving Usual Care; Test type: Superiority; p = 0.44, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Neonatal Intensive Care Unit Admission
Description: Number of neonates admitted to the neonatal intensive care unit for > 24 hours
Time Frame: Date of delivery to date of discharge from hospital, assessed up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 43 | 42
Participants | 15 | 21
Statistical Analysis 1: Comparison: Neonates Born to Mothers Receiving Intervention vs Neonates Born to Mothers Receiving Usual Care; Test type: Superiority; p = 0.16, Chi-squared

10. Secondary Outcome: Neonatal Intensive Care Unit Length of Stay
Description: Number of days of neonatal intensive care unit stay
Time Frame: From neonatal intensive care unit admission to discharge, assessed up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 43 | 42
days | 6 [4 to 13] | 7 [2 to 11]
Statistical Analysis 1: Comparison: Neonates Born to Mothers Receiving Intervention vs Neonates Born to Mothers Receiving Usual Care; Test type: Superiority; p = 0.59, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Neonatal Seizures
Description: Number of neonates who had seizures
Time Frame: After birth, during hospital admission, assessed up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 43 | 42
Participants | 0 | 0

12. Secondary Outcome: Neonatal Mortality
Description: Number of neonates who died
Time Frame: After birth, during hospital admission, assessed up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
Number analyzed (Participants) | 43 | 42
Participants | 0 | 0

13. Secondary Outcome: Maternal Hyperglycemia
Description: Number of mothers with intrapartum capillary blood glucose >110 mg/dL, fasting capillary blood glucose >95 mg/dL, or 1-hour postprandial capillary blood glucose >140 mg/dL
Time Frame: For five days after first dose of betamethasone administration
Population: Only 39 participants in the intervention group had at least one capillary blood glucose measured
Measure: Count of Participants; unit: Participants
Groups:
- Mothers: Intervention: Mothers will undergo regular maternal blood glucose screening and treatment of hyperglycemia following BMZ administration to achieve maternal glycemic control until delivery or hospital discharge, for a maximum of 5 days.
- Mothers: Usual Care: Routine antenatal care will be performed without any maternal blood glucose screening nor treatment as is usual care at each of the study sites.
Arm/Group | Mothers: Intervention | Mothers: Usual Care
Number analyzed (Participants) | 39 | 0
Participants | 32 | 0

14. Secondary Outcome: Maternal Insulin Treatment
Description: Number of mothers who received insulin for treatment of hyperglycemia
Time Frame: For five days after first dose of betamethasone administration
Population: Only 39 mothers in the intervention group had at least one capillary blood glucose measured
Measure: Count of Participants; unit: Participants
Arm/Group | Mothers: Intervention | Mothers: Usual Care
Number analyzed (Participants) | 39 | 0
Participants | 22 |

15. Secondary Outcome: Maternal Hypoglycemia
Description: Number of mothers with capillary blood glucose <60 mg/dL
Time Frame: For five days after first dose of betamethasone administration
Population: Only 39 mothers in the intervention group had at least one capillary blood glucose measured
Measure: Count of Participants; unit: Participants
Arm/Group | Mothers: Intervention | Mothers: Usual Care
Number analyzed (Participants) | 39 | 0
Participants | 0 |

ADVERSE EVENTS:
Time Frame: Collected for mothers from the time of informed consent until delivery or hospital discharge for a maximum of 5 days. For neonates, AEs were collected from the time of birth until discharge or 28 days of life.
Arm/Group | Mothers: Intervention | Mothers: Usual Care | Neonates Born to Mothers Receiving Intervention | Neonates Born to Mothers Receiving Usual Care
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/42 | 0/43 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/42 | 0/43 | 0/42
Other Adverse Events (participants affected / at risk) | 11/44 | 7/42 | 30/43 | 35/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Mothers: Intervention (N=44) | Mothers: Usual Care (N=42) | Neonates Born to Mothers Receiving Intervention (N=43) | Neonates Born to Mothers Receiving Usual Care (N=42)
Neonatal Hypoglycemia (Endocrine disorders) | 0/0 (0) | 0/0 (0) | 20 (20) | 21 (21)
Neonatal Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 6 (6) | 4 (4)
Transient Tachypnea of the Newborn (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 3 (3) | 2 (2)
Neonatal Apnea (Respiratory, thoracic and mediastinal disorders) | 0/0 (0) | 0/0 (0) | 2 (2) | 4 (4)
Neonatal Hyperbilirubinemia (Hepatobiliary disorders) | 0/0 (0) | 0/0 (0) | 10 (10) | 18 (18)
Cesarean delivery (Reproductive system and breast disorders) | 11/43 (11) | 7 (7) | 0/0 (0) | 0/0 (0)
Neonatal Intensive Care Unit Admission (General disorders) | 0/0 (0) | 0/0 (0) | 15 (15) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT03076775/Prot_SAP_000.pdf